CLINICAL TRIAL: NCT01905085
Title: Energy Expenditure Methodology Infant
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 133331
Record Dates: First submitted 2013-07-09; First posted 2013-07-23 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: No intervention

SUMMARY:
Indirect calorimetry is valuable in determining resting energy expenditure in infants, children and adults. This measure will estimate the number of calories needed per day under resting conditions.

Adding physical activity measures will help estimate total energy requirements in individuals. With the rise in obesity, numerous programs of prevention are being developed. Being able to characterize carefully energy intake and energy expenditure is one of the challenges of most of these initiatives.

ELIGIBILITY:
Inclusion Criteria:

* 3 months old +/- 2 weeks
* Can fall asleep easily
* Usually sleeps more than 30 min
* Accept formula as an alternative feeding

Exclusion Criteria:

* Pulmonary or respiratory disorders

Ages: 3 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Measure Resting energy expenditure in infants | 2 days
  We will measure resting energy expenditure in infants and then they will come back for a second visit and get the same measurement to see if there is a significant difference between the two measures.